CLINICAL TRIAL: NCT03173092
Title: An Open-Label, Single-Arm, Multicenter Study to Evaluate the Effectiveness and Safety of Ixazomib (NINLARO®) in Combination With Lenalidomide and Dexamethasone (IRD) in Patients With Multiple Myeloma Previously Receiving a Bortezomib-Based Induction Regimen (US MM-6)
Brief Title: A Study of Ixazomib (NINLARO®) in Combination With Lenalidomide and Dexamethasone (IRD) for the Treatment of Participants With Multiple Myeloma (MM)
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C16038; U1111-1192-7696 (Other: WHO)
Record Dates: First submitted 2017-05-30; First posted 2017-06-01 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Multiple Myeloma
Keywords: Drug therapy
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ixazomib 4 mg + Lenalidomide 25 mg + Dexamethasone 40 mg (Experimental): Ixazomib 4 milligram (mg), capsules, orally, once, on Days 1, 8 and 15 and lenalidomide 25 mg, capsules, orally, once on Days 1 through 21; and dexamethasone 40 mg, tablets, orally, once on Days 1, 8, 15 and 22 of a 28-day cycle for a maximum of 39 cycles until PD or unacceptable toxicity, whichever occurs first for up to 3 years.
  Interventions: Drug: Ixazomib; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Ixazomib — Ixazomib capsules.
  Other Names: NINLARO; MLN9708
Drug: Lenalidomide — Lenalidomide capsules.
Drug: Dexamethasone — Dexamethasone.

SUMMARY:
The main aim is to evaluate the effect of Ixazomib in combination with lenalidomide and dexamethasone on Multiple Myeloma disease progression at 2 years in participants who previously received a bortezomib-based induction regimen.

The study will enroll approximately 160 participants, who are enrolled after completing 3 cycles of chemotherapy (Bortezomib-Based Induction Regimen). They are then treated with Ixazomib in addition to lenalidomide and dexamethasone.

DETAILED DESCRIPTION:
The drug being tested in this study is called Ixazomib. Ixazomib is being tested to treat people who have MM. This study will look at the effectiveness and safety in participants who take the all-oral combination of ixazomib added to lenalidomide and dexamethasone.

The study will enroll approximately 160 participants. Participants will initially receive:

• Ixazomib 4 mg + lenalidomide 25 mg + dexamethasone 40 mg

Participants include MM participants who have received 3 cycles of a bortezomib-based induction regimen (as defined by current National Comprehensive Cancer Network [NCCN] guidelines) and have no evidence of PD following initial first-line therapy. All participants will be asked to take ixazomib 4 mg on Days 1, 8 and 15 and lenalidomide 25 mg from Day 1 through 21 and dexamethasone 40 mg on Days 1, 8, 15 and 22 in 28 day cycles until disease progression or unacceptable toxicity for up to 3 years.

Dose modifications of ixazomib, and/or lenalidomide and/or dexamethasone are allowed at the discretion of the physician.

This multi-center trial will be conducted in United States. It is anticipated that the treatment phase of this study will last up to 78 months, including 42 months for enrollment, and a 36-month IRD treatment period (39 cycles) with ixazomib and/or lenalidomide and/or dexamethasone for the last participant enrolled.

Participants will make multiple visits to the clinic as per their standard of care, and will be followed for PFS. After disease progression, participants will be followed-up for overall survival every 6 months until death or termination of the study by the sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Must have a diagnosis of a MM using current IMWG diagnostic criteria and have received 1 prior line of therapy.

   * Participants must have completed 3 cycles of a bortezomib-based induction regimen (as defined by current NCCN guidelines) and have no evidence of disease progression as defined by IMWG criteria.
   * Participants with light chain and free light chain (FLC) only may be enrolled if they meet all the criteria for a diagnosis of MM.
   * Participants must be considered by their physician eligible to receiving the IRD regimen.
2. Must be transplant ineligible as determined by their physician, or if transplant eligible, not expect to undergo transplant for at least 24 months after study enrollment.

   o Stem cell harvest and mobilization regimen is acceptable if clinically indicated, but must first be confirmed by the Takeda Medical Monitor.
3. Eastern Cooperative Oncology Group (ECOG) performance status and/or other performance status 0, 1, or 2 at time of enrollment.
4. Female participants who:

   * Are postmenopausal for at least 1 year before the screening visit, OR
   * Are surgically sterile, OR
   * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, OR
   * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the participant (periodic abstinence [example, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception).
5. Male participants, even if surgically sterilized (that is, status post-vasectomy), must agree to one of the following:

   * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
   * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence (example, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception).

Exclusion Criteria:

1. Participation in other interventional clinical trials, including those with other investigational agents not included in this trial, within 30 days of the start of this trial and throughout the duration of this trial. Non-interventional trials (that is, observational trials) are permitted at any time point.
2. Failure to have fully recovered (that is, less than or equal to [<=] Grade 1 toxicity) from the reversible effects of prior chemotherapy.
3. Major surgery within 14 days before enrollment.
4. Radiotherapy within 14 days before enrollment (if the involved field is small, 7 days will be considered a sufficient interval between treatment and administration of the ixazomib).
5. Central nervous system involvement by MM.
6. Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment.
7. Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months.
8. Systemic treatment, within 14 days before the first dose of ixazomib, with strong cytochrome P450 3A (CYP3A) inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort.
9. Ongoing or active systemic infection, active hepatitis B or C virus infection, or known human immunodeficiency virus positive.
10. Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Participants with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
11. Has greater than or equal to (>=) Grade 2 peripheral neuropathy, or Grade 1 with pain on clinical examination during the screening period.
12. Have previously been treated with ixazomib, or participated in a study with ixazomib whether treated with ixazomib or not.
13. PD on first-line therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | From date of first study drug administration until disease progression or death due to any cause, whichever occurs first (Up to 2 years).
  PFS is defined as time from date of first administration of study drug regimen to date of first documentation of progressive disease (PD) based on local laboratory results and investigator's assessment using modified International Myeloma Working Group (IMWG) response criteria or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Percentage of Participants with Partial Response (PR), Very Good Partial Response (VGPR) and Complete Response (CR) | Day 1 of each cycle (every 28 days) until disease progression for up to 3 years.
  Response is based on investigator's assessment using modified IMWG criteria.
Duration of Response | Day 1 of each cycle (every 28 days) until disease progression for up to 3 years.
  Duration of response is defined as the time from the date of first documentation of a PR or better to the date of first documentation of PD for responders.
Duration of Treatment (DoT) | From the date of the first study drug administration to the date of the last administration of any of the 3 study drugs (Up to 3 years).
  DoT is defined as the time from the date of the first administration of the study drug regimen (IRD) to the date of the last administration of any of the 3 study drugs in the regimen.
Duration of Ixazomib Therapy | From the date of the first ixazomib administration to the date of the last ixazomib administration (Up to 3 years).
  Duration of ixazomib therapy is defined as the time from the date of the first administration of ixazomib therapy to the date of the last administration of ixazomib therapy.
Relative Dose Intensity (RDI) for Each Study Drug | Up to 3 years
  RDI for each study drug is defined as 100*(Total amount of dose taken)/(Total prescribed dose of treated cycles), where total prescribed dose equals [dose prescribed at enrollment * number of prescribed doses per cycle * the number of treated cycles].
Duration of Proteasome Inhibitor Therapy | Up to 3 years.
  Duration of proteasome inhibitor therapy is defined as the time from the date of the first administration of bortezomib based therapy to the date of the last administration of the study drug (ixazomib).

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (21):
- United States (21):
  - Arizona Oncology Associates, Tucson, Arizona
  - Los Angeles Cancer Network/(Formerly -Pacific Cancer Medical Center), Anaheim, California
  - Compassionate Care Research Group, Inc., Fountain Valley, California
  - Innovative Clinical Research, Santa Ana, California
  - US Oncology Research, Colorado Springs, Colorado
  - Woodlands Medical Specialists- Pensacola, Pensacola, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Investigator Clinical Research - Indiana, Indianapolis, Indiana
  - Saint Agnes Hospital, Baltimore, Maryland
  - American Oncology Partners of Maryland P.A, Bethesda, Maryland
  - Central Care Cancer Center, Bolivar, Missouri
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - Comprehensive Cancer Center of Nevada, Henderson, Nevada
  - Tri-Health Cancer Institute-Medical Oncology and Hematology Westside, Cincinnati, Ohio
  - Willamette Valley Cancer Institute and Research Center - Springfield, Springfield, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Texas Oncology- Presbyterian Cancer Center Dallas, Dallas, Texas
  - Texas Oncology-San Antonio Northwest, San Antonio, Texas
  - Millennium Physicians Association, Shenandoah, Texas
  - Texas Oncology -Tyler, Tyler, Texas

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Rifkin RM, Costello CL, Birhiray RE, Kambhampati S, Richter J, Abonour R, Lee HC, Stokes M, Ren K, Stull DM, Cherepanov D, Bogard K, Noga SJ, Girnius S. In-class transition from bortezomib-based therapy to IRd is an effective approach in newly diagnosed multiple myeloma. Future Oncol. 2024 Jan;20(3):131-143. doi: 10.2217/fon-2023-0272. Epub 2023 Oct 9. PMID 37807952